CLINICAL TRIAL: NCT01378884
Title: Monitoring Study for the Use of Gastroparesis for Patient Who Have Failed Standard Therapy
Brief Title: The Use of Domperidone for Gastroparesis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Allegiance Health (Other)
Responsible Party: Ivan Cubas, MD, Allegiance Health Gastroenterology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH 10-001
Record Dates: First submitted 2010-02-03; First posted 2011-06-23 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Domperidone; Motilium
MeSH Terms: conditions — Gastroparesis | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Domeperidone (Experimental): Patients to receive Domperidone for treatment of Gastroparesis
  Interventions: Drug: Domperidone

INTERVENTIONS:
Drug: Domperidone — Patient to receive treatment with Domperidone
  Other Names: Domperidone / Motilium

SUMMARY:
The purpose of this study is to determine whether domperidone can be used safely and effectively for patient with gastroparesis.

DETAILED DESCRIPTION:
Individuals who have been diagnosed with gastroparesis and have failed at least one standard therapy will be offered to trial domperidone as a possible remedy to their condition. Patients on the medication will be expected to to be followed by the physician at 3 months, 6 months 12months, and then annually while on the medication. Any change or significant adverse reaction to the medication or in their condition should be reported immediately to their physician.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18 or older
3. Symptoms or manifestations secondary to GERD (e.g., persistent esophagitis, heartburn, upper airway signs or symptoms or respiratory symptoms), gastrointestinal motility disorders such as nausea, vomiting, severe dyspepsia or severe chronic constipation that are refractory to standard therapy.
4. Subjects must have a comprehensive evaluation to eliminate other causes of their symptoms.
5. Subject has signed informed consent for the administration of domperidone. The informed consent informs the subject of potential adverse events including:

   * increased prolactin levels,
   * extrapyramidal side effects,
   * breast changes,
   * cardiac arrhythmias including QT prolongation, and

Exclusion Criteria:

1. History of or current cardiac disease, including ischemic or valvular heart disease, other structural heart defects, cardiomyopathy or congestive heart failure.
2. History of or current arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsade des Pointes. Subjects with minor forms of ectopy (PACs) are not necessarily excluded.
3. Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QT syndrome (QTc greater than 450 milliseconds for males, greater 470 milliseconds for females) or family history prolonged QT syndrome.
4. Presence of a prolactinoma (prolactin-releasing pituitary tumor).
5. Conditions that result in electrolyte disorders, such as severe dehydration, vomiting, malnutrition, eating disorders, renal diseases, or the use of potassium-wasting diuretics or insulin in acute settings. (Note that the presence of vomiting, that may accompany gastroparesis or pseudo-obstruction does not by itself exclude the subject - only if accompanied by electrolyte disturbance must the subject be excluded.)
6. Pregnant or breast feeding female.
7. Known allergy to domperidone or any components of the domperidone formulation.
8. Significantly significant electrolyte disorders.
9. Gastrointestinal hemorrhage or obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Improved Gastric motility | 3 months
  Patients will have improved gastric motility within three months of begining domperidone therpy

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Cubas, MD, Principal Investigator — Allegiance Health Gastroenterology